CLINICAL TRIAL: NCT05907980
Title: A Phase Ia/Ib Open-label, Dose-escalation Study to Evaluate the Safety and Pharmacokinetics of ROSE12 as a Single Agent and in Combination With Other Anti-tumor Agents in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Phase I Study of ROSE12 Alone and in Combination With Other Anti-tumor Agents in Patients With Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RSE101CT
Record Dates: First submitted 2023-04-20; First posted 2023-06-18 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumor
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A: Dose-escalation part of Phase Ia (Experimental): Patients will receive ROSE12 as a IV infusion at escalated doses.
  Interventions: Drug: ROSE12
- Part B: Biopsy part of Phase Ia (Experimental): Serial biopsy will be conducted with patients who will receive ROSE12 as a IV infusion at escalated doses.
  Interventions: Drug: ROSE12
- Part C: Dose-escalation part of Phase Ib (Experimental): Patients will receive ROSE12 and atezolizumab as a IV infusion at escalated doses.
  Interventions: Drug: ROSE12; Drug: Atezolizumab
- Part D: Biopsy part of Phase Ib (Experimental): Serial biopsy will be conducted with patients who will receive ROSE12 and atezolizumab as a IV infusion at escalated doses.
  Interventions: Drug: ROSE12; Drug: Atezolizumab
- Part E: Expansion part of Phase Ib in patients with selected solid tumors (Experimental): Patients will receive ROSE12 and atezolizumab as a IV infusion at the recommended dose.
  Interventions: Drug: ROSE12; Drug: Atezolizumab

INTERVENTIONS:
Drug: ROSE12 — ROSE12 as a IV infusion
Drug: Atezolizumab — Atezolizumab as a IV infusion
  Arms: Part C: Dose-escalation part of Phase Ib; Part D: Biopsy part of Phase Ib; Part E: Expansion part of Phase Ib in patients with selected solid tumors

SUMMARY:
This is a Phase Ia/Ib open-label, dose-escalation study to evaluate the safety and pharmacokinetics of ROSE12 as a single agent and in combination with other anti-tumor agents in patients with locally advanced or metastatic solid tumors. The study will consist of three parts: a dose-escalation part, a biopsy part (the part to evaluate biomarkers), and an expansion part.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years at time of signing informed consent form (ICF)
* Eastern Cooperative Oncology Group (ECOG) PS of 0 or 1
* Adequate hematologic and end-organ function
* Life expectancy >= 12 weeks
* Patients with histologic documentation of locally advanced, or metastatic solid tumor
* [Dose-escalation Parts and Biopsy Parts]Refractory or resistant to standard therapies or standard therapies are not available
* [Dose-escalation Parts and Expansion Part] Patients with confirmed availability of fresh tumor or representative tumor specimens
* [Biopsy Parts] Patients with accessible lesion(s)

Exclusion Criteria:

* Clinically significant cardiovascular or liver disease
* Treatment with investigational therapy and anti-cancer therapy within 28 days prior to initiation of study drug
* Any history of an immune-mediated Grade 4 adverse event attributed to prior cancer immunotherapy (other than asymptomatic elevation of serum amylase or lipase).
* All imAEs from prior cancer immunotherapy (other than endocrinopathy managed with replacement therapy, stable vitiligo or stable alopecia) that have not resolved completely to baseline.
* Adverse events from prior anti-cancer therapy that have not resolved to Grade ≤ 1 except for alopecia, vitiligo, or endocrinopathy managed with replacement therapy
* Primary central nervous system (CNS) malignancy, untreated CNS metastases requiring any anti-tumor treatment, or active CNS metastases
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
* Active or history of clinically significant autoimmune disease
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.

[Expansion Part]

* Prior treatment with investigational product which has MoA of Treg depletion
* Malignancies other than disease under study within 5 years prior to Cycle 1 Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) and the recommended dose (RD) of ROSE12 when administered as a single agent and in combination with atezolizumab (Part A and C) | From Cycle 1 Day 1 until Cycle 1 Day 21 (Cycle 1 is 21 days)
  Incidence and nature of dose-limiting toxicities (DLTs)
Safety (All Parts) and tolerability (Part A, B, C and D) of ROSE12 when administered as a single agent and in combination with atezolizumab (Adverse Events) | From screening until study completion, treatment discontinuation or post-treatment follow up, assessed up to the end of the study (approximate 43 months)
  Incidence, nature, and severity of adverse events graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
The maximum serum concentration (Cmax) of ROSE12 for PK profile when administered as a single agent and in combination with atezolizumab (All Parts) | From Cycle 1 Day 1 (Cycle 1 is 21 days) until study completion or treatment discontinuation, assessed up to the end of the study (approximate 43 months)
  The maximum serum concentration (Cmax) of ROSE12
The minimum serum concentration (Cmin) of ROSE12 for PK profile when administered as a single agent and in combination with atezolizumab (All Parts) | From Cycle 1 Day 1 (Cycle 1 is 21 days) until study completion or treatment discontinuation, assessed up to the end of the study (approximate 43 months)
  The minimum serum concentration (Cmin) of ROSE12
The area under the concentration time-curve (AUC) of ROSE12 for PK profile when administered as a single agent and in combination with atezolizumab (All Parts) | From Cycle 1 Day 1 (Cycle 1 is 21 days) until study completion or treatment discontinuation, assessed up to the end of the study (approximate 43 months)
  The area under the concentration time-curve (AUC) of ROSE12
Preliminary anti-tumor activity of ROSE12 when administered in combination with atezolizumab (Part E) | From screening until study completion or treatment discontinuation, assessed up to the end of the study (approximate 43 months)
  Objective response rate (ORR), defined as the proportion of patients with an objective response (complete response [CR] or partial response [PR]) on two consecutive occasions ≥ 4 weeks apart, as determined by the investigator according to the Response Evaluation Criteria in Solid Tumors version 1.1

SECONDARY OUTCOMES:
Preliminary anti-tumor activity of ROSE12 when administered as a single agent and in combination with atezolizumab (Part A, B, C and D) | From screening until study completion or treatment discontinuation, assessed up to the end of the study (approximate 43 months)
  ORR, defined as the proportion of patients with an objective response on two consecutive occasions ≥ 4 weeks apart, as determined by the investigator according to RECIST v1.1.
Preliminary anti-tumor activity of ROSE12 when administered as a single agent and in combination with atezolizumab (All Parts) | From screening until study completion or treatment discontinuation, assessed up to the end of the study (approximate 43 months)
  Disease control rate (DCR), defined as the proportion of patients who had an objective response or stable disease (SD) which is confirmed no less than 6 weeks after the start of treatment as the minimum duration, as determined by the investigator with use of RECIST v1.1.
Preliminary anti-tumor activity of ROSE12 when administered as a single agent and in combination with atezolizumab (All Parts) | From screening until study completion or treatment discontinuation, assessed up to the end of the study (approximate 43 months)
  Duration of objective response (DoR), defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1.
Preliminary anti-tumor activity of ROSE12 when administered as a single agent and in combination with atezolizumab (All Parts) | From screening until study completion or treatment discontinuation, assessed up to the end of the study (approximate 43 months)
  Progression-free survival (PFS), defined as the time from administration of first study treatment to the first occurrence of disease progression or death from any cause, as determined by the investigator according to RECIST v1.1.
The maximum serum concentration (Cmax) of atezolizumab for PK profile when administered in combination with ROSE12 (Part C, D and E) | From Cycle 1 Day 1 (Cycle 1 is 21 days) until study completion or treatment discontinuation, assessed up to the end of the study (approximate 43 months)
  The maximum serum concentration (Cmax) of atezolizumab
The minimum serum concentration (Cmin) of atezolizumab for PK profile when administered in combination with ROSE12 (Part C, D and E) | From Cycle 1 Day 1 (Cycle 1 is 21 days) until study completion or treatment discontinuation, assessed up to the end of the study (approximate 43 months)
  The minimum serum concentration (Cmin) of atezolizumab
The area under the concentration-time curve (AUC) of atezolizumab for PK profile when administered in combination with ROSE12 (Part C, D and E) | From Cycle 1 Day 1 (Cycle 1 is 21 days) until study completion or treatment discontinuation, assessed up to the end of the study (approximate 43 months)
  The area under the concentration-time curve (AUC) of atezolizumab
The immunogenicity of ROSE12 when administered as a single agent and in combination with atezolizumab (All Parts) | From Cycle 1 Day 1 (Cycle 1 is 21 days) until study completion or treatment discontinuation, assessed up to the end of the study (approximate 43 months)
  Prevalence and incidence of anti-drug antibodies (ADAs) to ROSE12 and potential correlation with PK parameters and safety
The immunogenicity of atezolizumab when administered in combination with ROSE12 (Part C, D and E) | From Cycle 1 Day 1 (Cycle 1 is 21 days) until study completion or treatment discontinuation, assessed up to the end of the study (approximate 43 months)
  Prevalence and incidence of ADAs to atezolizumab and potential correlation with PK parameters and safety

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor Chugai Pharmaceutical Co.Ltd, Study Director — clinical-trials@chugai-pharm.co.jp
Locations (4):
- United States (2):
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, Fairfax, Virginia
- Japan (2):
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - National Cancer Center Hospital, Chuo-ku, Tokyo

REFERENCES:
- [Derived] Hayashi H, Tatsumi K, Katada H, Matsuda Y, Tsunenari T, Honda M, Nemoto T, Shimizu S, Miura-Okuda M, Ikuta Y, Ito A, Ogami C, Kato C, Kamimura M, Kibayashi T, Kubo C, Komatsu S, Komori Y, Shinozuka J, Susumu H, Tanno H, Tomii Y, Nakagawa K, Nagano H, Nanami M, Nishito Y, Fujisawa N, Matsushita T, Michisaka S, Yamazaki M, Yoshimoto M, Wakatsuki H, Wakabayashi T, Wada NA, Ueda O, Konishi H, Kashima K, Tanaka H, Endo M, Kitazawa T, Sakaguchi S, Kamata-Sakurai M, Igawa T. ROSE12, a novel anti-CTLA-4 FcgammaRs binding-enhanced antibody activated by extracellular adenosine triphosphate, shows tumor-selective regulatory T-cell depletion and antitumor efficacy without systemic immune activation. J Immunother Cancer. 2026 Jan 9;14(1):e013397. doi: 10.1136/jitc-2025-013397. PMID 41513409